CLINICAL TRIAL: NCT03026504
Title: Baricitinib in Relapsing Giant Cell Arteritis (GCA): A Phase II, Single-institution, Open-label Pilot Study
Brief Title: Baricitinib in Relapsing Giant Cell Arteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew J Koster (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor-Investigator, Matthew J Koster, MD, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-008993
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Arteritis, Giant Cell
MeSH Terms: conditions — Giant Cell Arteritis | interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Baricitinib Therapy (Experimental): 4 milligrams oral Baricitinib daily for 52 weeks
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — 4 milligrams oral Baricitinib daily for 52 weeks
  Other Names: JAK2 Inhibitor

SUMMARY:
This study will evaluate the safety and effectiveness of baricitinib in the treatment of giant cell arteritis. All participants will be taking prednisone at the start of the study. The prednisone will be reduced according to a standardized tapering schedule while participants continue to take one tablet of baricitinib daily for 52 weeks.

DETAILED DESCRIPTION:
Baricitinib, an orally administered, potent, selective and reversible inhibitor of JAK1 and JAK2 has shown preliminary safety and efficacy in chronic, immune-mediated inflammatory conditions such as rheumatoid arthritis and psoriasis. This small molecule is uniquely suited as a potential novel therapeutic agent in GCA because of its suppressive effect on both the Th17 (IL-6, IL-23) andTh1 (IL-12, IFN-γ) pathways.

This study will evaluate the safety and tolerability of baricitinib in a population of patients with relapsing GCA. The study is an open-label pilot study assessing the safety and tolerability of baricitinib (4 mg daily, oral, for 52 weeks) in addition to a standardized glucocorticoid taper. It is anticipated that adjunct baricitinib will be safe and well tolerated by patients with GCA and demonstrate preliminary efficacy as measured by reducing inflammatory markers, decreasing steroid requirements and increasing relapse-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Giant Cell Arteritis (GCA) defined by the following Revised GCA Diagnosis Criteria:

   * Age ≥50 years.
   * History of Erythrocyte Sedimentation Rate (ESR) ≥ 50 mm/hour or C-Reactive Protein (CRP) ≥ 10 mg/L.
   * Presence of at least one of the following:

     * Unequivocal cranial symptoms of GCA (new onset localized headache, scalp or temporal artery tenderness, otherwise unexplained mouth or jaw pain upon mastication).
     * Unequivocal symptoms of Polymyalgia Rheumatica (PMR), defined as shoulder and/or hip girdle pain associated with inflammatory stiffness.
     * Systemic inflammatory disease in which the presence of the fever (>38 degrees Celsius for ≥ 7 days), weight loss (> 5 pounds or 10% premorbid weight), and/or night sweats were attributable to GCA and no other cause was identified.
   * Presence of at least one of the following:

     * Temporal artery biopsy revealing features of GCA.
     * Evidence of large-vessel vasculitis by angiography or cross-sectional imaging, including but not limited to magnetic resonance angiography (MRA), computed tomography angiography (CTA), positron emission tomography-computed tomography (PET-CT) or evidence of large-vessel or temporal artery vasculitis by ultrasound (US).
2. Relapse with active GCA within 6 weeks of study entry where active disease is defined by an ESR ≥30 mm/hr or CRP ≥10 mg/L AND the presence of at least one of the following:

   * Unequivocal cranial symptoms of GCA (new onset or recurrent localized headache, scalp or temporal artery tenderness, otherwise unexplained mouth or jaw pain upon mastication [i.e., jaw claudication]).
   * Unequivocal symptoms of PMR, defined as shoulder and/or hip girdle pain associated with inflammatory stiffness.
   * Other feature(s) judged by the clinician investigator to be consistent with GCA or PMR flares (e.g. fever of unknown origin, weight loss, fatigue/malaise, etc.)
3. Clinically stable at baseline visit (study drug initiation) such that the subject is able to safely participate in the standardized taper regimen in the opinion of the investigator.

Exclusion Criteria

1. Presence of any other autoimmune disease (such as systemic lupus erythematosus, rheumatoid arthritis, inflammatory arthritis, other vasculitides, scleroderma, polymyositis, dermatomyositis, or other similar systemic connective tissue diseases).
2. Subjects demonstrating symptoms of visual loss (transient or permanent blindness) or diplopia attributable to GCA.
3. Subjects with history of aortic dissection, myocardial infarction, or cerebrovascular attack attributable to GCA.
4. Has received, or is expected to receive, any live virus vaccinations (with the exception of herpes zoster vaccination) within 3 months before the first dose of study drug, during the study, or within 3 months after the last administration of the study drug. All patients who have not received the herpes zoster vaccine at screening will be encouraged (per local guidelines) to do so prior to randomization; vaccination must occur >4 weeks prior to randomization and start of investigational product. Patients will be excluded if they were exposed to herpes zoster vaccination within 4 weeks of planned randomization.
5. Organ transplant recipients.
6. Have had a major surgery within 8 weeks prior to screening or will require major surgery during the study that, in the opinion of the investigator would pose an unacceptable risk to the patient.
7. Have experienced any of the following within 12 weeks of screening: myocardial infarction (MI), unstable ischemic heart disease, stroke, or New York Heart Association Stage IV heart failure
8. Have a history or presence of cardiovascular (including but not limited to uncontrolled hypertension), respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders, or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking investigational product or interfere with the interpretation of data.
9. Are largely or wholly incapacitated permitting little or no self-care, such as being bedridden or confined to a wheelchair.
10. Have an estimated glomerular filtration rate (eGFR) of <50 mL/min/1.73 m^².
11. Have a history of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2 times the upper limit of normal (ULN) or the most recent available total bilirubin ≥1.5 times ULN (if available).
12. Have a history of lymphoproliferative disease; or have signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or have active primary or recurrent malignant disease; or have been in remission from clinically significant malignancy for < 5 years.

    1. Subjects with uterine cervical carcinoma in situ that has been resected with no evidence of recurrence or metastatic disease for at least 3 years may participate in the study
    2. Subjects with basal cell or squamous epithelial skin cancers which have been completely resected with no evidence of recurrence for at least 3 years may participate in the study.
13. Active infections, or history of recurrent infections or have required management of acute or chronic infections as evidenced by any of the following:

    1. Currently on any suppressive therapy for a chronic infection (such as tuberculosis, cytomegalovirus, herpes simplex, herpes zoster, or atypical mycobacteria).
    2. History or suspicion of chronic infection (e.g. prosthetic joint infection)
    3. Hospitalization for treatment of infection within 60 days of baseline visit
    4. Use of parenteral (IV or IM) antimicrobials (antibacterial, antifungals, antivirals, or antiparasitic agents) within 60 days of baseline or oral antimicrobials within 30 days of baseline visit for treatment of an active infection. This does not include the use of antibiotics for prophylaxis against pneumocystis pneumonia since this is considered standard of care for patients on prednisone ≥ 20 mg/day for longer than 3 consecutive months.
14. Have had symptomatic herpes zoster infection within 12 weeks prior to screening.
15. Have a history of disseminated/complicated herpes zoster [for example, multidermatomal involvement, ophthalmic zoster or Central Nervous System (CNS) involvement]
16. In the opinion of the investigator, are at an unacceptable risk for participating in the study.
17. Have known or documented diagnosis of human immunodeficiency virus (HIV).
18. Have known or documented primary immunodeficiency.
19. Have had household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB.
20. Have had evidence of active TB or have previously had evidence of active TB and did not receive appropriate and documented treatment.
21. Have evidence of latent TB as documented by a local lab positive QuantiFERON®-TB Gold test and a normal chest x-ray, unless a patient completes at least 4 weeks of appropriate treatment prior to study entry and agrees to complete the remainder of treatment while in the trial.

    1. If the QuantiFERON®-TB Gold test results are positive, the patient will be considered to have latent TB and will be excluded. If the test is indeterminate, the test may be repeated once within 2 weeks of the initial value. If the repeat test results are again not negative, the subject will be considered to have latent TB (for purposes of this study) and will be excluded.
    2. Exceptions include subjects with a history of active or latent TB who have documented evidence of appropriate treatment and with no history of re-exposure since their treatment was completed. (Such subjects would not be required to undergo the protocol specific TB testing, but would require a baseline chest x-ray).
22. Have a positive test for Hepatitis B Virus (HBV) defined as:

    1. Positive for hepatitis B surface antigen (HBsAg), or
    2. Positive for anti-hepatitis B core antibody (HBcAb) If any of the Hepatitis B tests have an indeterminate result, confirmatory testing will be performed by an alternate method.
23. Have Hepatitis C Virus (HCV) (positive for anti-hepatitis C antibody with confirmed presence of HCV).
24. Have any of the following specific abnormalities on screening tests:

    1. ALT or AST > 2 x ULN
    2. Total bilirubin ≥1.5 x ULN
    3. Hemoglobin < 10 grams/deciliter
    4. Total white blood cell count (WBC) < 2500 cells/μL)
    5. Neutropenia (absolute neutrophil count [ANC] < 1200 cells/μL
    6. Lymphopenia (lymphocyte count < 750 cells/μL)
    7. Thrombocytopenia (platelets < 100,000 cells/μL)
    8. eGFR < 50 mL/min/1.73m²

    In the case of any of the aforementioned laboratory abnormalities, the tests may be repeated once within approximately 2 weeks from the initial values, and values resulting from repeat testing may be accepted for enrollment eligibility if they meet the eligibility criterion.
25. Are pregnant or breast feeding at the time of screening or enrollment.
26. Are females of childbearing potential who do not agree to use 2 forms of highly effective birth control when engaging in sexual intercourse with a male partner while enrolled in the study and for at least 4 weeks following the last dose of the study drug

    1. Females of non-childbearing potential are defined as women ≥60 years of age, women

       ≥40 but <60 years of age what had had cessation of menses for at least 12 months, or whom who are congenitally or surgically sterile (that is have had a hysterectomy, or bilateral oophorectomy or tubal ligation)
    2. The following birth control methods are considered highly effective (the subject should choose 2 to be used with their male partner

    i. Oral, injectable, or implanted hormonal contraceptives ii. Condom with spermicidal foam, gel film, cream or suppository iii. Occlusive cap (diaphragm or cervical/vault caps) with a spermicidal foam, gel, film, cream or suppository iv. . Intrauterine device v. Intrauterine system (for example progestin-releasing coil) vi. Vasectomies male (with appropriate post-vasectomy documentation of the absence of sperm in the ejaculate)
27. Are males who do not agree to use 2 forms of highly effective birth control (see above) while engaging in sexual intercourse with females partners of childbearing potential while enrolled in the study and for 4 weeks after the last dose of the study drug.
28. Have donated more than a single unit of blood within 4 weeks prior to screening or intend to donate blood during the course of the study.
29. Have a history of chronic alcohol abuse, IV drug abuse, or other illicit drug above within the 2 years prior to screening.
30. Have previously received baricitinib for other investigational study.
31. Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures
32. Are currently enrolled in, or discontinued within 4 weeks prior to screening from any other clinical trial involving an investigational product or nonapproved use of a drug or device or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
33. Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling whether biological or legally adopted.
34. Have a chronic medical illness requiring the use of oral of IV glucocorticoid treatment (e.g. asthma or emphysema) during the trial or requiring long term glucocorticoid treatment such that they would not be able to safely undergone a standardized glucocorticoid taper.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Warrington, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koster MJ, Crowson CS, Giblon RE, Jaquith JM, Duarte-Garcia A, Matteson EL, Weyand CM, Warrington KJ. Baricitinib for relapsing giant cell arteritis: a prospective open-label 52-week pilot study. Ann Rheum Dis. 2022 Jun;81(6):861-867. doi: 10.1136/annrheumdis-2021-221961. Epub 2022 Feb 21. PMID 35190385
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: All participants assigned to baricitinib 4 mg daily orally for 52 weeks.
Period: Overall Study
Arm/Group | Single Arm
Started | 15
Completed | 14
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Baricitinib Therapy
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Duration of GCA [Median (Inter-Quartile Range); unit: months] | 9 [7 to 21]
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.3 (3.4)
Median number of prior GCA relapses [Median (Full Range); unit: events] | 1 [1 to 2]
Baseline Predinose dose [Count of Participants; unit: Participants]
  30 mg/day | 4
  20 mg/day | 6
  10 mg/day | 5

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: The percentage of subjects who experienced greater than or equal to one adverse event
Time Frame: 52 weeks
Measure: Number; unit: percentage of subjects
Arm/Group | Baricitinib Therapy
Number analyzed (Participants) | 15
percentage of subjects | 93

2. Secondary Outcome: Giant Cell Arteritis (GCA) Relapse
Description: The number of subjects to experience relapse of GCA at 24 weeks and 52 weeks. As defined as:
  Presence of ESR ≥30 mm/hour and/or CRP ≥10 mg/L and the presence of at least one of the following:
  * Unequivocal cranial symptoms of GCA.
  * Unequivocal symptoms of PMR.
  * Other features judged by the clinician to be consistent with GCA or PMR (eg, fever of unknown origin, unexplained weight loss, fatigue/ malaise, etc) for which no other aetiology was identified as causational.
Time Frame: 24 weeks, 52 weeks
Population: One subject withdrawn at week 8. Data was not collected or analyzed for week 24 and week 52
Measure: Count of Participants; unit: Participants
Arm/Group | Baricitinib Therapy
Number analyzed (Participants) | 14
Participants
  24 Weeks | 1
  52 Weeks | 1

3. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR)
Description: ESR is a blood test that detects and monitors inflammation in the body. The normal range is 0 to 22 mm/hr for men and 0 to 29 mm/hr for women.
Time Frame: week 0, week 24, week 52
Population: One subject withdrawn at week 8. Data was not collected or analyzed for week 24 and week 52
Measure: Median (Inter-Quartile Range); unit: mm/hr
Arm/Group | Baricitinib Therapy
Number analyzed (Participants) | 15
mm/hr
  Week 0 | 7 [6 to 17]
  Week 24: number analyzed (Participants) | 14
  Week 24 | 13 [7 to 19]
  Week 52: number analyzed (Participants) | 14
  Week 52 | 10 [5 to 17]

4. Secondary Outcome: C Reactive Protein (CRP)
Description: C-reactive protein is a substance produced by the liver in response to inflammation. Normal blood CRP levels are below 3.0 mg/L.
Time Frame: week 0, week 24, week 52
Population: One subject withdrawn at week 8. Data was not collected or analyzed for week 24 and week 52. NA indicates CRP levels are < 3 mg/L, but lab values do not return any actual values that are below this level of detection. Unable to use the "<" symbol.
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Baricitinib Therapy
Number analyzed (Participants) | 15
mg/L
  Week 0 | 3.4 [NA to 6.9] — N/A indicates CRP levels are < 3 mg/L, but lab values do not return any actual values that are below this level of detection. Unable to use the "<" symbol.
  Week 24: number analyzed (Participants) | 14
  Week 24 | NA [NA to NA] — N/A indicates CRP levels are < 3 mg/L, but lab values do not return any actual values that are below this level of detection. Unable to use the "<" symbol.
  Week 52: number analyzed (Participants) | 14
  Week 52 | NA [NA to 3.1] — N/A indicates CRP levels are < 3 mg/L, but lab values do not return any actual values that are below this level of detection. Unable to use the "<" symbol.

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately 64 weeks.
Arm/Group | Baricitinib Therapy
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baricitinib Therapy (N=15)
thrombocytopenia (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Baricitinib Therapy (N=15)
Infection not requiring antibiotics (Infections and infestations) | 8
Infection requiring antibiotics (Infections and infestations) | 5
Nausea (Gastrointestinal disorders) | 6
Edema limbs - leg (General disorders) | 2
Fatigue (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03026504/Prot_SAP_000.pdf